CLINICAL TRIAL: NCT01793792
Title: Pivotal Study of the Microvention, Inc Neurovascular Self-Expanding Retrievable Stent System LVIS
Brief Title: Pivotal Study of the LVIS (Low Profile Visualized Intraluminal Support)
Acronym: LVIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL11002; G110188/S004 (Other: FDA)
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2019-11

CONDITIONS: Intracranial Aneurysms
Keywords: intracranial, saccular, aneurysms, stenting, coiling
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Intervention Model Description: Low Profile Visualized Intraluminal Support device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device: LVIS (Other): The LVIS Device is intended for use with embolization coils for the treatment of wide neck, intracranial aneurysms.
  Device: LVIS™ and LVIS™ Jr. MicroVention Low-profile Visualized Intraluminal Support Device
  Interventions: Device: LVIS™ and LVIS™ Jr

INTERVENTIONS:
Device: LVIS™ and LVIS™ Jr — The LVIS Device is intended for use with embolization coils for the treatment of wide neck, intracranial aneurysms.
  Other Names: Low Profile Visualized Intraluminal Support device

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Low Profile Visualized Intraluminal Support(LVIS™ and LVIS™ Jr.)devices from MicroVention, Inc. when used to facilitate endovascular coiling of wide-necked intracranial aneurysms with coils.

ELIGIBILITY:
Inclusion Criteria:

* Subject age between 18 and 75 years
* Subject with an unruptured or ruptured(>30days since occurence), wide-necked (neck ≥4mm or dome to neck ratio <2)intracranial saccular aneurysm (<20mm maximum diameter in any plane)

Exclusion Criteria:

* Subject with significant extra or intracranial stenosis of the parent artery (>50%) proximal to the target aneurysm.
* Subject with any condition which in the opinion of the treating physician would place the subject at high risk of embolic stroke
* Subject with contraindications to the use of antiplatelet agents
* Subject who is unable to complete the required follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2013-07; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Fiorella, M.D., Principal Investigator — Stony Brook University Medical Center
Locations (21):
- United States (21):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Dignity Health/Mercy San Juan Medical Center, Carmichael, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Health and Hospital, Oak Lawn, Illinois
  - Indiana University/Methodist Research Institute, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Albany Medical College, Albany, New York
  - University at Buffalo Neurosurgery, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - The Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Fiorella D, Boulos A, Turk AS, Siddiqui AH, Arthur AS, Diaz O, Lopes DK; LVIS investigators. The safety and effectiveness of the LVIS stent system for the treatment of wide-necked cerebral aneurysms: final results of the pivotal US LVIS trial. J Neurointerv Surg. 2019 Apr;11(4):357-361. doi: 10.1136/neurintsurg-2018-014309. Epub 2018 Oct 8. PMID 30297543
- See also: The safety and effectiveness of the LVIS stent system for the treatment of wide-necked cerebral aneurysms: final results of the pivotal US LVIS trial. Fiorella D, Boulos A, Turk AS, Siddiqui AH, Arthur AS, Diaz O, Lopes DK on behalf of LVIS Investigators — https://jnis.bmj.com/content/early/2018/10/15/neurintsurg-2018-014309

RESULTS

PARTICIPANT FLOW:
Groups:
- Device: LVIS: Device: LVIS™ and LVIS™ Jr. MicroVention Low-profile Visualized Intraluminal Support Device
Period: Overall Study
Arm/Group | Device: LVIS
Started | 153 (153 treated: 1 attempted no device implanted, 152 device implanted.)
Treated | 153 (153 Treated, 152 implanted with device, 1 attempted no device implanted)
Completed | 141
Not Completed | 12
Not completed — Death | 5
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 1
Not completed — Device Not Implanted | 1

BASELINE CHARACTERISTICS:
Arm/Group | Device: LVIS
Number analyzed (Participants) | 153
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 123
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Composite Success "Number of Participants With Primary Effectiveness Composite Success (100% Aneurysm Occlusion Without Clinically Significant In-stent Stenosis or Target Aneurysm Retreatment"
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Device: LVIS
Number analyzed (Participants) | 153
Participants | 108

2. Primary Outcome: Primary Safety Composite Rate (Disabling Stroke With mRS Score Greater Than or Equal to 3, or Neurological Death Within 12 Months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Device: LVIS
Number analyzed (Participants) | 153
Participants | 9

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Device: LVIS
All-Cause Mortality (participants affected / at risk) | 6/153
Serious Adverse Events (participants affected / at risk) | 48/153
Other Adverse Events (participants affected / at risk) | 15/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: LVIS (N=153)
Aneurysm rupture (Nervous system disorders) | 4 (4)
Aphasia (Nervous system disorders) | 1 (1)
Dissection or perforation of the parent artery (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Intra-Parenchymal Hemorrhage (IPH) (Nervous system disorders) | 4 (4)
Neurological deficits (Nervous system disorders) | 3 (3)
Seizure (Nervous system disorders) | 3 (4)
Stent Thrombosis (Nervous system disorders) | 5 (5)
Stroke (Nervous system disorders) | 9 (11)
Sub-Arachnoid Hemorrhage (SAH) (Nervous system disorders) | 3 (3)
Sub-Dural Hematoma (SDH) (Nervous system disorders) | 3 (3)
TIA (Transient Ischemic Attack) (Nervous system disorders) | 5 (5)
Target aneurysm retreatment (Surgical and medical procedures) | 5 (5)
Thromboembolic event (Nervous system disorders) | 1 (1)
Vasospasm (Nervous system disorders) | 7 (7)
Visual impairment (Eye disorders) | 4 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: LVIS (N=153)
Headache (Nervous system disorders) | 15 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No